CLINICAL TRIAL: NCT01076491
Title: A Pilot Study to Investigate the Feasibility and Tolerability of Inhaling a High Dose of Dry Powder Mannitol (IDPM) Per Breath Administered Via a Dry Powder Inhaler Loaded With a Single Capsule in Subjects With Bronchiectasis
Brief Title: High Dose Inhaled Mannitol Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Dr Brett Charlton, Pharmaxis
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: DPM-DEV-102b; DPM-DEV-102b (Other: Pharmaxis Ltd)
Record Dates: First submitted 2009-11-11; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mannitol — inhaled mannitol - single doses of either 70 mg or 90 mg

SUMMARY:
This study is to investigate the safety and tolerability of high doses of inhaled mannitol in subjects with bronchiectasis to further direct development of an improved drug delivery system.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects with non-CF bronchiectasis
* FEV1 > 50 % predicted and > 1.0L

Exclusion Criteria:

* bronchiectasis due to CF or endobronchial lesion
* respiratory infection requiring IV antibiotics in last 4 weeks
* pregnancy
* significant haemoptysis in last 6 months
* active TB
* end stage ILD
* contraindications as determined by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
emitted dose | single measure

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia